CLINICAL TRIAL: NCT01541527
Title: Prevalence and Epitope Specificity of Non-neutralizing Antibodies in Haemophilia A Patients Without Inhibitors, Immunogenicity of B Domain: A Prospective Study
Brief Title: Non Neutralizing Antibodies: Prevalence and Characterization
Status: Withdrawn | Type: Observational
Why Stopped: Promoter's change
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hôpital de la Timone (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); University Hospital, Toulouse (Other); Centre Hospitalier Universitaire de Nice (Other); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: UF 8844
Record Dates: First submitted 2012-02-17; First posted 2012-03-01 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2012-02

CONDITIONS: Hemophilia A
Keywords: non neutralizing antibody; Epitopic profile; Clinical relevance
MeSH Terms: conditions — Hemophilia A | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe, moderate and mild HA patients: one Arm: biological collection of 300 severe, moderate and mild HA patients
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — One blood test entering in the usual follow-up of the patient

SUMMARY:
Antibodies (Abs) directed against factorVIII (FVIII) remain the main iatrogenic complication in haemophilia A (HA) patients. Anti-FVIII Abs inhibiting pro-coagulant properties of the molecule are named inhibitors whereas Abs directed towards non-functional epitopes are named non-neutralizing antibodies (NNA). These NNA are poorly studied and their prevalence is ill-defined.

In a recent retrospective study the investigators evaluated, in a cohort of 210 patients without inhibitor, the NNA prevalence and the NNA epitope specificity against the heavy chain (HC)or the light chain(LC). For the first time, the investigators used two x-MAP based assays: the first to determine the specificity of anti-FVIII Abs against the HC or the LC, the second to display Abs directed towards the B domain. NNA were found in 38 out of 210 patients (18).

Among this NNA positive population, 74% and 13% of patients had anti-FVIII Abs against both chains. The proportion of NNA directed towards the B domain was 18%.

Considering an approximate inhibitor prevalence of 30% and a NNA prevalence of 19% in severe HA patients, approximately 50% of severe HA patients develop an immune response against infused FVIII. Due to their unclear relevance, the NNA detection does not yet belong to the routine clinical practice.

However, in 2006, Dimichele advancedf a hypothesis concerning the influence of NNA on the variations in the kinectics of FVIII observed in certain patients.

The mechanism explaining the role of these NNA in the FVIII in the FVIII kinectics has not still been demonstrated.

The investigators propose to perform a multicentre prospective study with the aim to confirm, in severe, moderate and mild HA treated patietns, the NNA prevalence observed in our retrospective study, to study the evolution over time of the epitopemapping of these NNA and to explore the correlation between these NNA and clinical/biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* male with Age > 6 years
* Severe, moderate or mild treated HA patients with negative inhibitor titer (<0.6UB)
* An information form will be presented to the patient or his/her legal representative by the physician who includes the patient in the study protocol
* Patient with national insurance

Exclusion Criteria:

* Patient without his agreement for this study
* Patient deprived of freedom
* Patient without national insurance

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: severe, moderate and mild HA patients (sex: Male and age > 6 years)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
NNA prevalence | 18 months
  The primary outcome is the study of the development of ANN anti-FVIII at the severe, moderate or mild HA patients to establish prevalency of ACs targeted against the heavy chain, the light chain and the domains of the FVIII (6 months after the inclusion.
  The investigators will evaluate the NNA prevalence by the x-MAP technology.

SECONDARY OUTCOMES:
Relationship between clinical and biological parameters and NNA presence | 18 months
  The secondary outcomes assess the evolution in time of these Acs of isotypes IgG and the relationship between clinical and biological parameters (FVIII%, recovery,..) and NNA presence.
  The investigators will evaluate the secondary outcomes by the x-MAP technology.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier- Centre administratif André Benech, Montpellier, France

REFERENCES:
- [Result] Lavigne-Lissalde G, Rothschild C, Pouplard C, Lapalud P, Gruel Y, Schved JF, Granier C. Characteristics, mechanisms of action, and epitope mapping of anti-factor VIII antibodies. Clin Rev Allergy Immunol. 2009 Oct;37(2):67-79. doi: 10.1007/s12016-009-8119-0. PMID 19172415
- [Result] Lavigne-Lissalde G, Tarrade C, Lapalud P, Chtourou S, Schved JF, Granier C, Villard-Saussine S. Simultaneous detection and epitope mapping of anti-factor VIII antibodies. Thromb Haemost. 2008 Jun;99(6):1090-6. doi: 10.1160/TH07-08-0497. PMID 18521513
- [Result] Lavigne-Lissalde G, Lacroix-Desmazes S, Wootla B, Tarrade C, Schved JF, Kaveri SV, Granier C, Villard-Saussine S. Molecular characterization of human B domain-specific anti-factor VIII monoclonal antibodies generated in transgenic mice. Thromb Haemost. 2007 Jul;98(1):138-47. PMID 17598006